CLINICAL TRIAL: NCT04724642
Title: Efficacy and Safety of COVID-19 Vaccine in Patients After Allogeneic Hamatopoietic Cell Transplantation, CAR-T Therapy and With Primary Immune Deficiency - a Post Marketing Prospective Cohort Study
Brief Title: COVID-19 Vaccine in Patients After Allogeneic HCT, CAR-T Therapy and With Primary Immune Deficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1067-20
Record Dates: First submitted 2021-01-24; First posted 2021-01-26 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Allogenic Hematopoietic Cell Transplant; CAR-T Therapy; Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The corona pandemic is a continuing global challenge due to Corona Virus 2019 (COVID-19).

The purpose of the study is to confirm the accepted hypothesis from the recommendations of The European Society for Blood and Marrow Transplantation, that the vaccine for COVID-19 is safe and has good efficacy in immunocompromised patients after a bone marrow transplant from a donor / cellular therapy.

DETAILED DESCRIPTION:
The study population will be allogeneic bone marrow transplant patients and those who have received CART therapy - immunocompromised patients who are vaccinated with COVID-19 in a commercial preparation, regardless of the study.

The following procedures are routinely performed before receiving the vaccine in the bone marrow transplant unit -

1. Blood count and lymphocyte subgroup counts before vaccination (up to 48 hours before vaccination).
2. Evaluation of GVHD activity and accompanying toxicity.
3. Receipt of a letter confirming the vaccination to the HMO.
4. One-week follow-up after vaccination including blood count, complete chemistry, GVHD evaluation, and review of adverse reactions that may be vaccine-related.
5. Referral for a second dose of the vaccine.
6. One week follow-up after vaccination including blood count, complete chemistry, GVHD evaluation, review of side effects that may be vaccine related.

The following procedures are performed only as part of the study -

1. Serology test (IgG AntiS) two weeks after the second dose of the vaccine to test the effectiveness of the vaccine.

   Cell separation two weeks after the second vaccination and execution -
2. ELISpot test to test for the release of interferon gamma in response to the stimulation of cells separated with the SARS-COV-2 virus peptides (stimulation with S peptides to evaluate vaccine response, and stimulation with M peptides as a control).

All data collected in the study will be typed into Excel and analyzed using SPSS version 25.0. Continuous data will be described using averages and standard deviations, and categorical data will be described using prevalence and percentages.

The distribution of the continuous variables will be presented using an outline graph and will be examined using the Kolmogorov Smirnov test.

An attempt will be made to perform subgroup analysis (depending on the frequency of the groups in the sample) for the patient group:

Patients after bone marrow transplantation with acute GVHD Patients after bone marrow transplantation with chronic GVHD Patients after bone marrow transplantation without immunosuppressive therapy Patients after Cell Therapy (CART) Patients lack primary immunization

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Patient sex - male and female
* Bone marrow transplant from a donor (sibling or unrelated) or after cell therapy (CART) at least 3 months before vaccination.
* Patients with primary immunodeficiency syndrome.
* Patients who are able to sign an informed consent form

Exclusion Criteria:

* Patients under 18 years of age
* Patients who are unable to give informed consent
* Patients with acute GVHD who require steroid therapy above 0.5 mg / kg or who have been diagnosed in the last month.
* Patients with chronic GVHD who require steroid therapy above 0.5 mg / kg
* Patients treated with rituximab / immunoglobulins / mesenchymal cells during the last month.
* Patients whose disease is not completely cured and receive dedicated treatment for the disease.
* Patients receiving maintenance treatment for the underlying disease (excluding TKIs such as sorfenib, midostaurin, guiltritinib or cranolinib).
* Patients who have previously had COVID19.
* Patients with severe allergy to one of the vaccine components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients after allogeneic bone marrow transplant or after CART therapy and 40 patients with a primary immunodeficiency.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-05-28 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of side effects in patients | 10 weeks counting since first vaccination is initiated.
  Incidence of side effects in patients post allogeneic bone marrow transplantation after COVID-19 vaccination

SECONDARY OUTCOMES:
Prevalence of severe adverse reactions | 10 weeks counting since first vaccination is initiated.
  1. Prevalence of severe adverse reactions (grade 3-4) in patients post allogeneic bone marrow transplantation after vaccination with COVID-19
  2. Percentage of patients with SEROCONVERSION to COVID-19 (IgG Anti S)
  3. Exacerbation rates in GVHD - Acute GVHD - Exacerbation of GVHD in at least one organ by at least one grade without continued improvement of GVHD in the other affected organs.
     Chronic GVHD - Exacerbation of GVHD in each of the organs involved.
  4. Infection with COVID19, according to a PCR test from a nasopharyngeal sample

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ram, Prof, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel